CLINICAL TRIAL: NCT07373977
Title: Comparison of Postoperative Pain After Pulpotomy Performed With Versus Without Dental Operating Microscope in Carious Mature Permanent Teeth : A Randomized Controlled Trial
Brief Title: Comparison of Postoperative Pain After Pulpotomy Performed With Versus Without Dental Operating Microscope in Carious Mature Permanent Teeth
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Sirawut Hiran-us, Associate Professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BBC 42/2025
Record Dates: First submitted 2026-01-21; First posted 2026-01-28 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Carious Exposure of Pulp
Keywords: Pulpotomy; Dental operating microscope; post-operative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Additional using of dental operating microscope in the procedure (Experimental): using of dental operating microscope in the procedure to improve the quality of treatment
  Interventions: Device: Using dental operating microscope
- Rountine pulpotomy (No Intervention): Rountine pulpotomy procedure without addition using of dental operating microscope

INTERVENTIONS:
Device: Using dental operating microscope — Using dental operating microscope additional to the procedure
  Arms: Additional using of dental operating microscope in the procedure

SUMMARY:
The goal of this [randomized clinical trials] is to investigate the effect of using dental operating microscope incorperated in full pulpotomy procedure in mature carious posterior teeth.

The main questions it aims to answer are:

investigate postoperative pain levels.

investigate the quality of life of patient after treatment.

If there is a comparison group: Researchers will compare the pulpotomy procedure with and without using dental operating microscope.

Participants will will be asked to do

* Pain evaluation with numerical rating scale
* OHIP 14 survey before and after treatment

DETAILED DESCRIPTION:
Study design and setting This study is a prospective, single-center, single-blinded, parallel-group, randomized controlled trial conducted at the Dental Department, Phaholponpayuhasena Hospital. All clinical procedures are performed by a single experienced endodontist.

Study participants Inclusion Criteria

* Healthy patients aged at least 18 years old with deep or extremely deep carious lesions in mature permanent teeth diagnose with symptomatic irreversible pulpitis. Diagnoses are confirmed using EPT and cold tests. Pulpal and periapical diagnoses are based on terminology from the American Association of Endodontists.
* Posterior teeth with moderate or severe pain according to The NRS (Numeric Rating Scale) According to this scale, the level of pain is documented in the range of 0-10 numerically and verbally as no pain (0), mild pain, non-disruptive to routine activities (1-3), moderate pain that interferes with daily life but no need analgesics intake (4-6) and severe pain that significantly disrupts normal activities requiring analgesic intervention (7-10).
* Teeth that response negatively to percussion and palpation tests.
* Teeth are restorable with direct composite restoration. Exclusion Criteria
* Teeth with subgingival caries and/or clinical attachment loss more than 3 mm and probing depth more than 4 mm.
* Negative responses to pulp sensibility tests, presence of sinus tracts, swelling, non-restorable crowns, immature roots, or no pulp exposure following complete caries removal in case of pre-operative diagnosis as asymptomatic irreversible pulpitis.
* Patients with systemic diseases involving bleeding disorders such as hemophilia, Von Willebrand disease, platelet disorders. And patients under taking all kind of anticoagulant and anti-platelet.
* Patients who had taken analgesics or anti-inflammatory drugs within the previous 24 hours. If necessary, record how many and dose that taken.
* Patients taking opioids.
* Known allergies to non-steroidal anti-inflammatory drugs (NSAIDs).
* Pregnant or lactating patients.
* Teeth with pulpal obliteration.
* Necrotic pulp is found after access opening
* Bleed cannot be stopped within 8 minutes after full pulpotomy Treatment procedure A comprehensive medical and dental history is taken before treatment. Preoperative data, including age, sex, tooth number, and pain intensity are recorded in a predesigned patient's chart. The severity of pain is measured using NRS 0-10. The treatment, the study design, alternative treatment modalities, potential benefits, risks, and follow-up protocol are explained to the qualifying patients and informed consent is obtained from the voluntary patients who are willing to participate in the study.

Sample size calculation The sample size calculation was based on a study by Kubra G. and Koray Y. 2025 using a G*Power v.3.1 (Heinrich Heine, Dusseldorf University, Dusseldorf Germany) with a 95% power, a 5% α error, and an effect size of 0.75. The minimum sample size was calculated to be 78. Considering patients lost to follow-up, a total of 82 teeth from different patients are included in this study. Randomization and masking Block randomization with variable 4 block sizes is used to generate a sequence of random numbers for allocating the patients equally into two study groups. Each random blocks are sealed in an opaque envelope which is opened at the beginning of the clinical trial by the operator. New block will be open after all the patient in the previous block was completed and repeat until the end of the clinical trials to ensure the equality of group distribution: The vital pulp therapy with and without magnification intervention groups.

Intervention All the treatment is carried out by a single operator. All the patients received a topical anesthesia before local anesthesia. An inferior alveolar nerve block (1.8 ml 2% Lidocaine with epinephrine 1:100,000)+buccal infiltration (1.7 ml 4% Articaine with epinephrine 1:100,000) for mandibular teeth, buccal infiltration (1.8 ml 2% Lidocaine with epinephrine 1:100,000) for maxillary teeth. The anesthesia is confirmed by negative response to EPT. The pulpotomy procedure is performed under rubber dam isolation in a single visit. If the patient experienced pain during the procedure, an additional anesthesia is used to achieve profound pulpal anesthesia by intraligament injection with 0.3 ml 2% Lidocaine with epinephrine 1:100,000. The operating field is disinfected with iodine and alcohol. .A cylindrical diamond airotor operates under air water coolant to outline the cavity. Low speed round bur and a spoon excavator are used to remove the soft carious dentine using nonselective caries removal from the periphery towards the centre of the carious lesion. The deepest layer of carious dentine is thereafter disinfected with 2 ml of 2.5% NaOCl prior to pulpal exposure.

The patient will have his or her eyes covered with a dental drape and randomly divided into the following two groups:

Group I (Magnification) : The remaining procedures will be carried on under Zeiss OPMI Pico dental operating microscope (Carl Zeiss Meditec, Germany) with total magnification ranging from 3.6× to 6.0×. More aspects will be included in this group which included:

* If the remaining resected pulp is avascular with necrotic or yellowish liquefied areas, or microscopic hemostasis cannot be achieved, then further tissue removal is attempted
* Ensure the absence of dentin chips and blood clotting above remaining pulp tissue.
* Complete removal of detached pulp tissue and dentine fragments into a vascular pulp.

Group II (Control) : The remaining procedures will be carried on under naked eye.

The new high-speed sterile diamond airotor is used to completely remove the coronal pulp tissue. Then direct passive irrigation with of 2.5% NaOCl solution up to 8 minutes to arrest the bleeding. The time to achieve hemostasis is recorded in minutes and seconds. The diagnosis of vital inflamed pulp is confirmed by the presence of bleeding in the pulp chamber.

In both study groups, 1 mm calcium silicate cement putty type (Totalfil-ERRM) is placed as a caping agent over the residual pulp. The tooth is restored with Resin Modified Glass Ionomer Cement (RMGIC) base (Vitrebond, 3M) and composite restoration (Z350XT, 3M) and polishing in the same visit.

The full pulpotomy cases where bleeding from residual pulp cannot be arrested within 8 minutes, are excluded from the study, and pulpectomy are performed. Immediate post-operative periapical radiograph is taken.

Post-operative evaluation The patient's postoperative pain score and frequency of analgesic intake are recorded during at 6, 24, 48, and 72-hours. Ibuprofen 400 mg 10 tablets and Paracetamol 500 mg 10 tablets will be prescribed for every patient in advance.

If patients have a complaint of pain, they can have 1 tablet of ibuprofen 400 mg, with a note down the number and time of intake.

If the patient can't tolerate the pain after taken 1 tablet of ibuprofen for 60 minutes, there can have another 1 tablet of paracetamol, with a note down the number and time of intake.

Patients are also informed to return to the clinician in case of persistent severe pain in the post-intervention period, even after taking prescribed medication.

Patient also be asked for doing OHIP-14 survey before and after treatment.

Statistical analysis The Kolmogorov-Smirnov test is used to assess the normality of continuous data. Fisher's exact test analyze demographic variables. Pain intensity and analgesic use are compared using the t-test or Mann- Whitney U test. Intra- and intergroup comparisons of pain intensity at different intervals are performed using the Wilcoxon signed-rank test. A p-value of < 0.05 is considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients aged at least 18 years old with deep or extremely deep carious lesions in mature permanent teeth diagnose with symptomatic irreversible pulpitis. Diagnoses are confirmed using EPT and cold tests. Pulpal and periapical diagnoses are based on terminology from the American Association of Endodontists (AAE, 2013)20.
* Posterior teeth with moderate or severe pain according to The NRS (Numeric Rating Scale) According to this scale, the level of pain is documented in the range of 0-10 numerically and verbally as no pain (0), mild pain, non-disruptive to routine activities (1-3), moderate pain that interferes with daily life but no need analgesics intake (4-6) and severe pain that significantly disrupts normal acitivities requiring analgesic intervention (7-10).
* Teeth that response negatively to percussion and palpation tests.
* Teeth are restorable with direct composite restoration.

Exclusion Criteria:

* Teeth with subgingival caries and/or clinical attachment loss more than 3 mm and probing depth more than 4 mm.
* Negative responses to pulp sensibility tests, presence of sinus tracts, swelling, non-restorable crowns, immature roots, or no pulp exposure following complete caries removal in case of pre-operative diagnosis as asymptomatic irreversible pulpitis.
* Patients with systemic diseases involving bleeding disorders such as hemophilia, Von Willebrand disease, platelet disorders. And patients under taking all kind of anticoagulant and anti-platelet.
* Patients who had taken analgesics or anti-inflammatory drugs within the previous 24 hours. If necessary, record how many and dose that taken.
* Patients taking opioids.
* Known allergies to non-steroidal anti-inflammatory drugs (NSAIDs).
* Pregnant or lactating patients.
* Teeth with pulpal obliteration.
* Necrotic pulp is found after access opening
* Bleed cannot be stopped within 8 minutes after full pulpotomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2026-02-10 (Estimated); Primary Completion 2026-12-28 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 72 hrs after treatment
  Patient will be asked to do a post-operative pain assessment by using numerical rating scale before and after treatment a 6hr, 24 hrs, 48 hrs, 72 hrs.
  Minimum is 0, Maximum is 10 Higher the score worsen the outcome.

SECONDARY OUTCOMES:
Patient's quality of life assessment | 72 hrs after treatment
  Patient will be asked to do OHIP-14 survey before and after treatment Minimum is 14, Maximum is 70 Higher the score worsen the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Sirawut Hiran-us, DDS, MSc, High Grad Dip, FRCDS, Study Director — Faculty of Dentistry, Chulalongkorn University; Choontawee Soponsakulkaew, DDS, Higher Grad Dip, FRCDS, Principal Investigator — Phaholpolpayuhasena Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chang Ya-Ching, Wang Ting-Ya, Effectiveness of microscope-assisted root canal treatment in permanent posterior teeth: A retrospective cohort study. Journal of Dentistry, 2025.157: 105771.